CLINICAL TRIAL: NCT06203886
Title: Exploratory Clinical Investigation of the LumbaCure® Medical Device Used in Elderly People Suffering From Chronic Low Back Pain.
Brief Title: Effect of the LumbaCure® Intervention on Elderly Patients Suffering From cLBP.
Acronym: LumbaCure2303
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-23-09-043961
Record Dates: First submitted 2023-12-13; First posted 2024-01-12 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Intervention arm (Experimental): LumbaCure robotic device
  Interventions: Device: LumbaCure

INTERVENTIONS:
Device: LumbaCure — LumbaCure® is a device developed to induce specific mobilization of the lower back in patients requiring physical rehabilitation for orthopaedic disorders, particularly chronic low back pain.

SUMMARY:
The goal of this investigation is to evaluate the safety and efficacy of the LumbaCure® device in elderly people suffering from low back pain. The study is being carried out at several sites, in nursing homes, in order to reach the elderly patients most at risk of a sedentary lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or sub-acute low back pain (without "red flag")
* The subject, a resident or worker at the investigation site (nursing home), over 60 years of age
* Ability to communicate with the physiotherapist.
* Ability to remain in a sitting position for at least 10 minutes.
* A level of back pain > 2 on the numerical pain rating scale

Exclusion Criteria:

* Suspected or confirmed serious pathology (infection, fracture, cancer, inflammatory arthritis, ....) related to the back/spine.
* Body weight > 120 kg
* Subject is non-ambulatory or has severely reduced mobility.
* Dominant component of radicular pain (common lumbago with distal radiation below the knee)
* Radiculopathy
* Severe cardiorespiratory disease
* Dementia or significant cognitive impairment that prevents the participant from giving consent, completing study questionnaires or complying with recommendations.
* Fracture or operation less than 3 months old of the spine, pelvis, hip or leg bones.
* Known vertebral pathology other than osteoarthritis.
* Major neurological disease, movement or motor neuron disorders
* Fibromyalgia or other systemic rheumatic disease
* Recent history of stroke or heart failure, unstable heart condition
* Uncontrolled substance abuse disorders
* Invasive procedures to relieve pain in the last 3 months
* Acute or terminal illness
* Any other medical condition considered by the study team to be a contraindication to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Low back pain | Change between baseline and Visit 3 (Day 28)
  Mean intensity of low back pain during the last week, assessed on a numerical pain rating scale from 0 to 10

SECONDARY OUTCOMES:
Functional mobility | Between baseline and visit 3 (day 28)
  Change in the time taken to complete the time up and go (TUG) test. The TUG consists of measuring the time it takes a person to get up from a chair, walk 3 metres at their usual pace, turn around, return to the chair and sit down. Two attempts are made and the best time is recorded
Functional mobility | Between baseline and visit 2 (Day 14)
  Change in the time taken to complete the time up and go (TUG) test. The TUG consists of measuring the time it takes a person to get up from a chair, walk 3 metres at their usual pace, turn around, return to the chair and sit down. Two attempts are made and the best time is recorded
Functional mobility | Follow-up period : between the end of the investigation period and 1 month post-study (Day 56 - Visit 4)
  Change in the time taken to complete the time up and go (TUG) test. The TUG consists of measuring the time it takes a person to get up from a chair, walk 3 metres at their usual pace, turn around, return to the chair and sit down. Two attempts are made and the best time is recorded
Low back pain | Between baseline and each week through study completion, one month.
  Weekly changes from baseline in mean intensity of low back pain during the last week, assessed on a numerical pain rating scale from 0 to 10.
Low back pain | Before and after each session [12 measures, 3x/week during one month]
  Current back pain intensity before and after each session, assessed on a numerical pain rating scale from 0 to 10.
Low back pain | Follow-up : Between end of the investigation period [Day 28] and 1 month post-study.
  Changes in mean intensity of low back pain in the last week, assessed on a numerical rating scale from 0 to 10, during the follow-up period between the end of the investigation period and 1 month post-study.
Overall satisfaction of the physiotherapist with the LumbaCure® intervention | End of intervention period [Day 28]
  A single satisfaction score will be reported at the end of the intervention period by the physiotherapist:
  * How satisfied or dissatisfied are you with the ability of the LumbaCure® device intervention to improve your patient's low back pain condition (7 point scale)?
  * To what extent are you satisfied or dissatisfied with the ability of the LumbaCure® device to improve your patient's mobilisation (7-point scale)?
Overall patient satisfaction with the LumbaCure® intervention | End of intervention period [Day 28]
  A single satisfaction score will be calculated at the end of the intervention period based on a series of three questions :
  * How satisfied or dissatisfied are you with the ability of the LumbaCure® procedure to improve your lower back pain (7 point scale)?
  * How satisfied or dissatisfied are you with the ability of the LumbaCure® procedure to improve your mobility?
  * How would you rate your overall experience with the LumbaCure® device (7-point scale)?
Risk of falling | Between baseline and the end of the investigation,visit 3 [Day 28]
  Change in the risk of falling between baseline and the end of the intervention period, visit 3 (day 28), assessed by the Tinetti test. This test is a comprehensive assessment of both balance and gait. It assesses the patient's ability to change position, maintain balance in different situations and walk.
Risk of falling | Between the end of the investigation,visit 3 [Day 28] and one month follow-up
  Changes in the risk of falling during the follow-up period assessed by the Tinetti test. This test is a comprehensive assessment of both balance and gait. It assesses the patient's ability to change position, maintain balance in different situations and walk.

OTHER OUTCOMES:
Safety of the device | through study completion, one month
  The number, intensity and severity of adverse events are reported before each LumbaCure session.

CONTACTS AND LOCATIONS:
Locations (1):
- ASBL " Mère Joséphine " - MRS Saint Joseph Blegny, Blégny, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No